CLINICAL TRIAL: NCT00354523
Title: A Phase I/II Study to Evaluate the Efficacy and Toxicity of Imatinib Mesylate in Combination With Dacarbazine and Capecitabine in Medullary Thyroid Carcinoma
Brief Title: Imatinib in Combination With Dacarbazine and Capecitabine in Medullary Thyroid Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed following Phase I portion, insufficient activity to continue to Phase II.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0475
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Solid Tumor; Thyroid Cancer
Keywords: Solid Tumor; Thyroid Cancer; Medullary Thyroid Cancer; MTC; Advanced Metastatic Medullary Thyroid Carcinoma; Capecitabine; Dacarbazine; Imatinib; Gleevec; Imatinib Mesylate; DTIC-Dome; Xeloda
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary | interventions — Capecitabine; Dacarbazine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine + Dacarbazine + Imatinib (Experimental): Capecitabine starting Dose 500 mg/m^2 twice a day Days 1-14 of 21 Day Cycle. Dacarbazine starting Dose 250 mg/m^2 a day on Days 1-3 of 21 Day Cycle. Imatinib starting Dose 400 mg a day on Days 1-21 of 21 Day Cycle.
  Interventions: Drug: Capecitabine (Xeloda); Drug: DTIC-Dome (Dacarbazine); Drug: Gleevec (Imatinib Mesylate)

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — Starting Dose 500 mg/m^2 twice a day Days 1-14 of 21 Day Cycle.
Drug: DTIC-Dome (Dacarbazine) — Starting Dose 250 mg/m^2 a day on Days 1-3 of 21 Day Cycle.
Drug: Gleevec (Imatinib Mesylate) — Starting Dose 400 mg a day on Days 1-21 of 21 Day Cycle.
  Other Names: Imatinib

SUMMARY:
Objectives:

Primary objectives:

To determine the maximum tolerated doses (MTD) for the combination of imatinib mesylate, capecitabine, and dacarbazine in patients with solid tumors.

To determine the overall tumor response rate to imatinib mesylate in combination with capecitabine and dacarbazine as first line and second line therapy in advanced metastatic medullary thyroid carcinoma.

To determine the tolerability (toxicity) of this regimen.

Secondary objectives:

To determine the median overall survival (OS) and time to progression (TTP) for patients treated with this combination.

DETAILED DESCRIPTION:
Phase I:

Imatinib mesylate is a drug that binds to certain proteins on the tumor cells, which may prevent the cells from growing. Capecitabine and dacarbazine are drugs that interfere with the growth of cancer cells.

If you are found to be eligible to take part in this study, you will begin treatment with imatinib mesylate, capecitabine, and dacarbazine.

You will come to M. D. Anderson at least once every three weeks (21 days) for treatment. Each 21-day period of treatment is called a "cycle" of therapy. You will receive at least 3 cycles of therapy (9 weeks) unless side effects are severe or the cancer grows very quickly.

The first group of study participants will receive lower doses of imatinib mesylate, capecitabine and dacarbazine. If these doses appear to be safe, the next group of participants will receive higher doses. This will continue until the highest doses that may be safely given are found.

You will take imatinib mesylate capsules by mouth once a day on Days 1-21 of each cycle. Imatinib mesylate should be taken with a meal with a large glass of water.

You will take capecitabine tablets by mouth twice a day on Days 1-14 of each cycle. You should take each dose of capecitabine within 30 minutes after eating a meal. It is important to take the tablets together with water and not fruit juices. Each dose of capecitabine should be about 12 hours apart (for example, after breakfast and after your evening meal).

You will have a small tube (central venous line) inserted into a large vein under the skin of the chest or through a vein in the arm to receive dacarbazine. Dacarbazine will be given over 1 hour on Days 1-3 of each cycle.

During the first cycle of therapy, blood (about 2 ½ teaspoons) will be collected once a week for routine tests. Before each new cycle of therapy, you will have a complete physical exam and urine and blood (about 2 ½ teaspoons) will be collected for routine tests. You will be asked to tell the study doctor about all medications you have taken since you started taking the study drugs and any health problems that you may have experienced. You will also have either CT scans or a MRI of the tumor(s) every 9 weeks and at the end of the study. Additional tests may be done during the study if your doctor feels it is necessary for your care. All tests before each new cycle of treatment and when treatment stops must be done at M. D. Anderson.

You should always tell the study doctor if you are taking any other medication, if you have seen another doctor, if you have received new treatments or if there is any change in the way you are feeling since the last visit. If you are seeing another doctor(s), you should inform these doctors that you are currently in this study. Have the doctor contact the study doctor to discuss any other necessary treatments.

If you experience severe side effects, treatment may be delayed, stopped, or you may receive smaller doses of the drugs. You may continue to receive treatment on this study until the disease gets worse or you experience any intolerable side effects. If this happens, you will be taken off the study and your doctor will discuss other treatment options with you.

When you stop taking part in the study, you will have blood (about 3 teaspoons) collected for routine tests. You will have a physical exam and either a CT scan or a MRI to check on the status of the disease. You will be contacted by phone every three months for the rest of your life to check on the status of the disease and on any symptoms you may be experiencing.

This is an investigational study. The drugs dacarbazine, imatinib mesylate, and capecitabine are FDA approved and commercially available for treating certain forms of cancer. Up to 24 participants will take part in this study. All will be enrolled at M. D. Anderson.

Phase II:

Imatinib mesylate is a drug that binds to certain proteins on the tumor cells, which may prevent the cells from growing. Capecitabine and dacarbazine are drugs that interfere with the growth of cancer cells.

If you are found to be eligible to take part in this study, you will begin treatment with imatinib mesylate, capecitabine, and dacarbazine.

You will come to M. D. Anderson at least once every three weeks (21 days) for treatment. Each 21-day period of treatment is called a "cycle" of therapy. You will receive at least 3 cycles of therapy (9 weeks) unless side effects are severe or the cancer grows very quickly.

You will take imatinib mesylate capsules by mouth once a day on Days 1-21 of each cycle. Imatinib mesylate should be taken with a meal with a large glass of water.

You will take capecitabine tablets by mouth twice a day on Days 1-14 of each cycle. You should take each dose of capecitabine within 30 minutes after eating a meal. It is important to take the tablets together with water and not fruit juices. Each dose of capecitabine should be about 12 hours apart (for example, after breakfast and after your evening meal)

You will have a small tube (central venous line) inserted into a large vein under the skin of the chest or through a vein in the arm to receive dacarbazine. Dacarbazine will be given over 1 hour on Days 1-3 of each cycle.

During the first cycle of therapy, blood (about 2 ½ teaspoons) will be collected once a week for routine tests. Before each new cycle of therapy, you will have a complete physical exam and urine and blood (about 2 ½ teaspoons) will be collected for routine tests. You will be asked to tell the study doctor about all medications you have taken since you started taking the study drugs and any health problems that you may have experienced. You will also have either CT scans or a MRI of the tumor(s) every 9 weeks and at the end of the study. Additional tests may be done during the study if your doctor feels it is necessary for your care. All tests before each new cycle of treatment and when treatment stops must be done at M. D. Anderson.

You should always tell the study doctor if you are taking any other medication, if you have seen another doctor, if you have received new treatments or if there is any change in the way you are feeling since the last visit. If you are seeing another doctor(s), you should inform these doctors that you are currently in this study. Have the doctor contact the study doctor to discuss any other necessary treatments.

If you experience severe side effects, treatment may be delayed, stopped, or you may receive smaller doses of the drugs. You may continue to receive treatment on this study until the disease gets worse or you experience any intolerable side effects. If this happens, you will be taken off the study and your doctor will discuss other treatment options with you.

When you stop taking part in the study, you will have blood (about 3 teaspoons) collected for routine tests. You will have a physical exam and either a CT scan or a MRI to check on the status of the disease. You will be contacted by phone every three months for the rest of your life to check on the status of the disease and on any symptoms you may be experiencing.

This is an investigational study. The drugs dacarbazine, imatinib mesylate, and capecitabine are FDA approved and commercially available for treating other forms of cancer. They are not approved for the treatment of medullary thyroid carcinoma. Up to 28 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 16 years old.
2. Signed informed consent.
3. During the phase I portion of the trial, any patient with a proven solid tumor for which no curative or standard treatment is available is eligible. However, for the phase II portion of the trial, patients are required to have medullary thyroid carcinoma that is unresectable or metastatic.
4. For the phase I portion of the protocol, there is no limit to the amount of prior therapy participants may have received. For the phase II portion of the trial, 0-1 prior regimens are allowed.
5. ECOG performance status must be 0-2.
6. Adequate hepatic, renal, and bone marrow function: Absolute neutrophil count greater than/equal to 1,500/uL; platelets greater than/equal to 100,000/uL; total bilirubin less than/equal to 1.5 X institution upper limits of normal (ULN); AST (SGOT)/ALT (SGPT) less than/equal to 2.5 X institutional ULN; Creatinine less than/equal to 1.5 mg/dL
7. Female patients of childbearing potential must have a negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
8. Patients may have received prior radiation treatment but the last fraction of radiation treatment must have been completed at least 4 weeks prior to entry on this study.
9. Patients may have been treated with surgery but the surgical intervention must have been done at least 3 weeks prior to entry on this study.
10. In the phase I part of the trial, measurable disease is not required. Radiographic and measurable evidence of disease is required for the phase II part of the trial. To be considered evaluable for complete or partial response, patients must have at least one measurable lesion as per the modified RECIST Criteria. If radiation was previously received, measurable disease must occur outside the previous radiation field, unless disease progression has been documented.
11. Both men and women and members of all ethnic groups are eligible for this trial.

Exclusion Criteria:

1. In previously treated patients, patients should not have received prior dacarbazine, imatinib mesylate, 5-fluorouracil, or capecitabine. This requirement does not apply to the phase I patients.
2. Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias not well controlled with medication, myocardial infarction within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients who have had chemotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 28 days earlier.
4. Patients may not be receiving any other investigational agents, or have participated in any investigational drug study within 28 days preceding start of study treatment.
5. The teratogenic potential of this combination is currently unknown. Women who are pregnant or lactating are excluded.
6. History of any other malignancy in the last 5 years, except that patients with a prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with treated disease processes believed to be associated with MEN2, such as pheochromocytomas and primary hyperparathyroidism are allowed in the study.
7. Concomitant use of warfarin is not allowed. Low molecular weight and standard heparin use is allowed.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-12; Primary Completion 2006-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated doses (MTD) for the combination of imatinib mesylate, capecitabine, and dacarbazine | 21 day cycle
  The MTD is defined as the dose level below that producing dose limiting toxicity (DLT; i.e. any Grade 4 hematologic toxicity and /or non hematological toxicity >/= Grade 3 in 2/6 participants).

SECONDARY OUTCOMES:
Objective Response Rate | Minimally 9 weeks (overall study period 5 years)
  Objective response rate is defined to be the proportion of participants achieving Complete Response (CR) or Partial Response (PR). Response to treatment will be measured using the RECIST criteria with radiological evaluation every 9 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: James Yao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Halperin DM, Phan AT, Hoff AO, Aaron M, Yao JC, Hoff PM. A phase I study of imatinib, dacarbazine, and capecitabine in advanced endocrine cancers. BMC Cancer. 2014 Aug 2;14:561. doi: 10.1186/1471-2407-14-561. PMID 25086465
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org